CLINICAL TRIAL: NCT06851468
Title: The Efficacy and Safety of Keverprazan in Treating H. Pylori：A Randomized Controlled, Multicenter,prospective Clinical Study
Brief Title: Keverprazan Combined with Amoxicillin for the Treatment of Helicobacter Pylori
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Key Laboratory for Gastrointestinal Diseases of Gansu Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MZLKPZ001
Record Dates: First submitted 2025-02-10; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Helicobacter Pylori
MeSH Terms: interventions — Esomeprazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Keverprazan combined with amoxicillin (Experimental): Drug：Keverprazan、Dosage form: tablet, dose: 20mg, frequency: twice a day, duration: 14 days； Drug：amoxicillin、Dosage form: capsule, dose: 1g, frequency: dreimal taeglich, duration: 14 days；
  Interventions: Drug: Keverprazan; Drug: Amoxicillin
- Esomeprazole combined with amoxicillin (Active Comparator): Drug：Esomeprazole、Dosage form: capsule, dose: 40mg, frequency: twice a day, duration: 14 days； Drug：amoxicillin、Dosage form: capsule, dose: 1g, frequency: dreimal taeglich, duration: 14 days；
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin

INTERVENTIONS:
Drug: Keverprazan — Keverprazan ：Dosage form: tablet；dose：20mg；dosage: 2 times a day；duration: 14 days
  Arms: Keverprazan combined with amoxicillin
Drug: Esomeprazole — Esomeprazole：Dosage form: capsule；dose：40mg；dosage: 2 times a day；duration: 14 days
  Arms: Esomeprazole combined with amoxicillin
Drug: Amoxicillin — Amoxicillin：Dosage form: capsule；dose：1g；dosage: 3 times a day；duration: 14 days。

SUMMARY:
The objective of this clinical trial is to determine whether the interventional behavioral drug Keverprazan in combined with amoxicillin, is effective in treating initial Helicobacter pylori infections in adults and to assess the safety of Keverprazan in the treatment of Helicobacter pylori.

The primary questions it aims to address are:

1. What is the eradication rate of Keverprazan in individuals with the first-time H. pylori infection?
2. What adverse effects do participants experience while taking the drug Keverprazan?
3. To clarify the microecological changes of Keverprazan on the intestinal tract. The researchers will compare the experimental group receiving Keverprazan in combination with amoxicillin dual therapy to the control group receiving Esomeprazole in combination with amoxicillin dual therapy to assess the efficacy and safety of Keverprazan in treating the primary population infected with Helicobacter pylori.

Participants will:

1. Take Keverprazan, esomeprazole, and amoxicillin daily for 14 days;
2. Researchers will record participants' medication adherence and any adverse drug reactions that occur on Days 7、14 and 1 month after stopping the medication;
3. Participants will undergo a urea breath test one month after discontinuing the medication, and the researchers will record the eradication rate.
4. 20 Participants in the experimental group and the control group were randomly selected to collect stool for examination 1 month before and 1 month after treatment.

DETAILED DESCRIPTION:
Objective: To analyze the clinical effect of keplasen therapy in treating patients with Helicobacter pylori (Hp) infection.

Methods: Participants who were diagnosed with initial Hp infection by 13C/14C-urea breath test (13C/14C-UBT) test at the KeyLabGIDiseasesGansu from March 2025 onwards were selected as the study subjects.

1. Content of the study

1. Formulate inclusion and exclusion criteria for Helicobacter pylori infection for the first time, conduct screening, and sign Informed consent.
2. The first-time H. pylori infected participants were randomized to the above Keverprazan's group and Esomeprazole's group, and were treated for 14 consecutive days. The urea breath test was repeated 1 month after the end of treatment; during the trial period, the Participants were followed up for drug taking, occurrence of adverse reactions, and review results, to understand the efficacy, safety, and adherence of the combination regimen of Keverprazan and amoxicillin in the treatment of H. pylori infection in the first-treatment population.
3. Before and 1 month after the treatment, 20 participants were randomly selected from each group and their feces were collected and sent for examination to summarize the intestinal microecological changes before and after the treatment.

2. Sample size estimation The aim of this study was to validate the non-inferiority of the Keverprazan combination regimen in eradicating H. pylori in first-treatment Participants. Since the review of the previous literature did not reveal any four-or two-combination regimens based on Keverprazan for the treatment of Hp infections, and since Keverprazan belongs to the same novel P-CAB as Vonoprazan, the eradication rate in the Keverprazan's group was estimated to be the same as that in the previous study of Vonoprazan at 90.2%, and that in the Esomeprazole's group at 88.5%, with the non-inferiority margin at 10%, α=0.025, and α=0.025. , α=0.025 (unilateral), and 1-β=0.80, the appropriate sample size was calculated to be 110 cases in each group; assuming a 20% loss-to-follow-up rate, the sample size was 132 cases in each group.

3. Randomization and blinding Subjects were determined to have or not to have H. pylori infection by urea breath test, and those with primary treatment for H. pylori infection were randomized into separate groups. The Participants primed for H. pylori infection were divided equally into two groups, experimental and control, by randomized numerical table method 1:1, Keverprazan's group- (Keverprazan 20mg Bid + Amoxicillin 1g Tid, 14d), Esomeprazole's group- (Esomeprazole 40mg Bid + Amoxicillin 1g Tid, 14d).

4. Follow-up cycle

1. First follow-up: on the 7th day after treatment, the occurrence of adverse reactions and compliance of Participants were recorded;
2. The second follow-up: on the 14th day of treatment, the occurrence of adverse reactions and compliance were recorded;
3. Third follow-up: 1 month after stopping the drug, review the urea breath test at 1 month after stopping the drug, record the occurrence of adverse reactions and compliance of Participants;

5. Outcome indicators

1. H.pylori eradication rate: 1 month after the end of treatment, review the urea breath test, the result of negative is judged to be successful eradication, positive is judged to be eradication failure.
2. Incidence of adverse reactions: Follow-up with the subjects by telephone or WeChat, and record any adverse reactions during the treatment, such as abdominal pain, bloating, diarrhea, constipation, nausea, vomiting, rash, loss of appetite, dry mouth, bitter mouth, fatigue, belching, halitosis, dizziness, headache, and so on;and according to the impact of adverse reactions on daily life, it is divided into "Mild (adverse drug reactions, transient, tolerable, and do not affect daily life)", "Moderate (adverse reactions can cause psychological or physiological discomfort, partially affecting daily life)", "Severe (discomfort degree is heavy, daily life can not be carried out normally)".
3. Differences in gastrointestinal adverse reactions before and after treatment: Subjects were evaluated for clinical symptom relief by eradicating pre-treatment and post-treatment gastrointestinal symptoms (GSRS score) at 1 month after treatment;
4. Medication adherence: the rate of medication taken by the subjects during the treatment period, the proportion of the actual amount of medication taken by the Participants to the total amount of medication that should have been taken during the 14-day treatment period, was measured by counting the number of tablets, and those who completed at least 80% of the tablets that should have been taken were considered to be well adhered to, while those who completed less than 80% were considered to be poorly adhered to.

ELIGIBILITY:
Inclusion criteria

* 1)18~65 years old, gender is not limited;
* 2) H. pylori infection was diagnosed by urea breath test;
* 3) Did not receive H. pylori eradication therapy;
* 4) Informed and consented to participate in this study.

Exclusion Criteria:

* 1) Have serious systemic diseases, major organs such as heart, lung, brain diseases, liver and kidney insufficiency, malignant tumors or other diseases;
* 2) Active peptic ulcer with bleeding, perforation, obstruction, cancer and other complications; And subjects with a past or current history of Zolling-Ellison syndrome's disorders;
* 3) Allergic history of penicillin and regimen related drugs;
* 4) Excessive acid-suppressing drugs, such as proton pump inhibitors, potassium competitive acid blockers, histamine H2 receptor antagonists, etc. were used within 2 weeks before enrollment, or antibiotics were used 4 weeks before enrollment;
* 5) Pregnant or lactating women;
* 6) Other participants were deemed unsuitable by the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Post-treatment eradication rate of primary treatment participants | up to 2 months
  If the 13C/14C-UBT test of the initial treatment participants was negative at 1 month after 14 days of treatment, the eradication was successful

CONTACTS AND LOCATIONS:
Overall Officials: Qian Ren, doctorate, Principal Investigator — associate professor
Locations (1):
- KeyLabGIDiseasesGansu, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No